CLINICAL TRIAL: NCT06401317
Title: Comparison of the Efficacy of Intra-Articular Corticosteroid Injections Versus Saline Solution for Thumb Osteoarthritis: Double-Blind Pragmatic Randomized Pilot Study
Brief Title: Corticosteroid Against Saline Injections for Thumb Osteoarthritis (CASITOA)
Acronym: CASITOA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other); McGill University (Other); Université de Montréal (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Principal Investigator, Tokiko Hamasaki, Assistant Professor, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASITOA
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Trapeziometacarpal Osteoarthritis
Keywords: Corticosteroids; Feasibility; Blinding; Randomized controlled trial; Saline; Trapeziometacarpal osteoarthritis; Intra-articular injection; Pragmatic trial
MeSH Terms: interventions — Saline Solution; Triamcinolone Acetonide; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: 2-arm pragmatic randomized controlled pilot trial
Who Masked: Participant, Care Provider
Masking Description: Participants will be randomly assigned in a 1:1 ratio to receive either the saline injection or the corticosteroid injection. Opaque syringes will be used to mask the content to both participants and clinicians. The study will use computer-generated randomization to prepare and distribute sealed, opaque envelopes. These envelopes, indicating whether saline or corticosteroids should be injected, will be randomly sent to the healthcare facilities of the doctors involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline Injection (Experimental): A single injection of saline solution
  Interventions: Drug: Saline Solution (NaCl 0,9%)
- Corticosteroid Injection (Active Comparator): Usual care, consisting on a single injection of corticosteroids
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Saline Solution (NaCl 0,9%) — Ultrasound/fluoroscopy-guided intra-articular injection of 0.25ml of 0.9% saline solution.
  Other Names: Saline solution
  Arms: Saline Injection
Drug: Triamcinolone Acetonide — Ultrasound-guided intra-articular injection 0.25ml (10 mg) of triamcinolone.
  Other Names: Corticosteroid
  Arms: Corticosteroid Injection

SUMMARY:
Thumb osteoarthritis or trapeziometacarpal osteoarthritis (TMO) is a common and painful form of hand arthritis that limits thumb mobility and hand function, affecting patients' quality of life. Although corticosteroids injections are a typical treatment, their effectiveness has been challenged, and side effects have been reported. Recent studies suggest that saline injections, usually considered inactive, might be a viable treatment option. The primary goal of this study is to compare the effectiveness of saline injections versus corticosteroids injections in reducing TMO-related pain and improving hand function. In this study, 40 people with TMO will be randomly assigned to receive either a corticosteroids or a saline injection, without them or the doctors performing the injection knowing which one was administered (double blind). If saline injections prove more effective, they could provide a less harmful and cheaper therapeutic alternative for TMO patients.

DETAILED DESCRIPTION:
Trapeziometacarpal osteoarthritis (TMO) is one of the most painful, disabling and prevalent hand osteoarthritis. One of the most common treatments for TMO is an intra-articular corticosteroids injection. However, non-superiority of corticosteroids injection over placebo to reduce pain has also been reported for TMO and other types of osteoarthritis (knee, hip, or shoulder). Furthermore, adverse effects of corticosteroids injection such as subcutaneous atrophy, tendon ruptures, and articular cartilage damage have been reported. Given the uncertain relevance of corticosteroids injection as a therapeutic agent, it becomes imperative to consider alternative options. In fact, three systematic reviews suggest that saline injections may be a viable option for TMO or knee pain.

To investigate the hypothesis that saline injection is a more effective modality than corticosteroids injection for the treatment of TMO in terms of reducing TMO pain and improving hand function, we must undertake a large, randomized trial in real clinical settings to ensure the acquisition of high-quality evidence. This pilot project is a preparatory phase for a larger study aimed at comparing the effectiveness of saline and corticosteroids injections in treating TMO, focusing on pain reduction and functional improvements. The study design is a pragmatic, double-blind randomized trial, adhering to PRECIS-2 guidelines.

The pilot randomized controlled trial will assess the feasibility of a study by evaluating aspects such as recruitment capabilities, treatment adherence, and the success of blinding techniques for participants and clinicians. It will also identify potential challenges and gather preliminary data to support a funding application for the full-scale study. Recruitment and data collection are planned over a 12-month period, targeting 40 participants initially to refine procedures and validate the study's feasibility. Participants will be randomly assigned to treatment, and the clinicians delivering the intervention will be blinded to the content of the injections. The study's primary outcome will measure pain intensity using a numeric scale at multiple time points, while secondary outcomes include upper limb functional limitations using the QuickDASH scale. These will be measured at baseline, before treatment, and at follow-up, 1, 3, and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years;
* diagnosis of TMO was confirmed by X-ray interpreted by a radiologist;
* suffering from pain at the base of the thumb;
* the attending physician deems that an intra-articular corticosteroid injection would be beneficial, rather than opting for other types of intervention such as surgery
* can read, understand and answer in either French or English.

Exclusion Criteria:

* having received one or more corticosteroid injections in the last 12 months or surgery on the affected thumb;
* suffering from painful thumb caused by a trauma (e.g., fracture, sprain), rheumatoid arthritis, or De Quervain's tendonitis; and
* being pregnant or breastfeeding; and
* known allergies to any components of the solutions (triamcinolone acetonide, benzyl alcohol, carboxymethylcellulose sodium, hydrochloric acid, polysorbate, sodium chloride, or sodium hydroxide) or to iodinated contrast media.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of participant recruitment | Through study completion (estimated time, 1 year)
  The number of participants recruited per week, raw and divided by those screened for eligibility and those deemed eligible
Rate of participants completing the follow-ups | Through study completion (estimated time, 1 year)
  The number of participants completing the follow-ups at 1, 3, and 6 months, divided by those recruited
Success of blinded procedures for clinicians | Up to 24 hours after each injection
  Success of blinded procedures for physicians will be by asking them by email after the injection to guess which treatment they administered. Three response categories for treatment guess: 'corticosteroid injection', 'saline injection', or 'I don't know'.
Success of blinded procedures for patients | 1, 3, and 6 months after receiving the injection
  Success of blinded procedures for patients will be investigated by asking them to guess which treatment they will have received via the post-injection questionnaire. Three response categories for treatment guess are 'corticosteroid injection', 'saline injection', or 'I don't know', after the last follow-up).

SECONDARY OUTCOMES:
Trapeziometacarpal pain intensity | Baseline, 1, 3, and 6 months after injection
  Three types of pain intensity (current, on the average in the last 7 days, at its worst in the last 7 days) will be measured using a 0-10 rating scale (0 = no pain and 10 = worst pain possible)
QuickDASH questionnaire (short version of the 30-item Disabilities of the Arm, Shoulder and Hand). | Baseline, 1, 3, and 6 months after injection
  11-item questionnaire assesses the level of physical function and symptoms among patients with upper limb musculoskeletal condition. The total score ranges from 0 to 100 and the higher it is, the more disabled is the patient.
Concomitant analgesic use | Baseline, 1, 3, and 6 months after injection
  This will be captured using the Cumulative Analgesic Consumption Score (CACS), a tool that combines a qualitative assessment based on the World Health Organization analgesic ladder with a quantitative evaluation based on a score computed from the number of analgesics taken from each of three different categories: acetaminophen/NSAIDs, weak opioids, and strong opioids.
Adverse events | 24 hours after the injection and at 1-month, 3-month- and 6-month post-injection.
  Side effects will be reported systematically by using a questionnaire with 5 items assessing the presence, type, frequency, severity and duration of injection-related adverse events.

OTHER OUTCOMES:
Second injection | 1, 3, and 6 months after injection
  The number of participants requesting a second injection with a different solution due to a perceived lack of efficacy, as well as the number of participants requesting a second injection with the same solution due to pain relapse will be compared between groups will be compared between groups (saline vs. cortisone)
Arthroplasty | 1, 3, and 6 months after injection
  The number of participants undergoing arthroplasty during the study period will also be compared between groups..

CONTACTS AND LOCATIONS:
Overall Officials: Tokiko Hamasaki, PhD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (2):
- Canada (2):
  - Centre Hospitalier de l'Université de Montréal - Physiatry, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal - Chirurgie plastique, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared by the investigators upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Undecided yet
Access Criteria: IPD will be shared by the investigators upon reasonable request

REFERENCES:
- [Background] Hansen PA, Roberts KB. Human situations: a course introducing physiology to medical students. Am J Physiol. 1991 Dec;261(6 Pt 3):S7-11. doi: 10.1152/advances.1991.261.6.S7. PMID 1755481
- [Background] Hamasaki T, Laprise S, Harris PG, Bureau NJ, Gaudreault N, Ziegler D, Choiniere M. Efficacy of Nonsurgical Interventions for Trapeziometacarpal (Thumb Base) Osteoarthritis: A Systematic Review. Arthritis Care Res (Hoboken). 2020 Dec;72(12):1719-1735. doi: 10.1002/acr.24084. Epub 2020 Nov 7. PMID 31600038
- [Background] Hamasaki T, Choiniere M, Harris PG, Bureau NJ, Gaudreault N, Patenaude N. Biopsychosocial factors associated with pain severity and hand disability in trapeziometacarpal osteoarthritis and non-surgical management. J Hand Ther. 2023 Jul-Sep;36(3):647-657. doi: 10.1016/j.jht.2022.10.001. Epub 2023 Mar 12. PMID 36918308
- [Background] Altman RD, Devji T, Bhandari M, Fierlinger A, Niazi F, Christensen R. Clinical benefit of intra-articular saline as a comparator in clinical trials of knee osteoarthritis treatments: A systematic review and meta-analysis of randomized trials. Semin Arthritis Rheum. 2016 Oct;46(2):151-159. doi: 10.1016/j.semarthrit.2016.04.003. Epub 2016 Apr 27. PMID 27238876
- [Background] Ayub S, Kaur J, Hui M, Espahbodi S, Hall M, Doherty M, Zhang W. Efficacy and safety of multiple intra-articular corticosteroid injections for osteoarthritis-a systematic review and meta-analysis of randomized controlled trials and observational studies. Rheumatology (Oxford). 2021 Apr 6;60(4):1629-1639. doi: 10.1093/rheumatology/keaa808. PMID 33432345
- [Background] Saltzman BM, Leroux T, Meyer MA, Basques BA, Chahal J, Bach BR Jr, Yanke AB, Cole BJ. The Therapeutic Effect of Intra-articular Normal Saline Injections for Knee Osteoarthritis: A Meta-analysis of Evidence Level 1 Studies. Am J Sports Med. 2017 Sep;45(11):2647-2653. doi: 10.1177/0363546516680607. Epub 2016 Dec 27. PMID 28027657
- [Background] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159
- [Background] Kirkeby OJ, Fossum S, Risoe C. Anaemia in elderly patients. Incidence and causes of low haemoglobin concentration in a city general practice. Scand J Prim Health Care. 1991 Sep;9(3):167-71. doi: 10.3109/02813439109018513. PMID 1754748